CLINICAL TRIAL: NCT00632450
Title: EnSite Real-Time Cardiac Performance Measurements Study, a Non-significant Risk Study
Brief Title: EnSite Real-Time Cardiac Performance Measurements (RT CPM) Study
Acronym: EnSite RT CPM
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 40004879
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
The EnSite Real-Time Cardiac Performance Measurements Study (EnSite RT CPM) is a multicenter, international, acute, non-significant risk study, designed to enroll a maximum of 40 patient. The goal of the study is to collect 3-D systolic/diastolic data with the EnSite NavX Mapping system during a CRT implant.

Patients enrolled in this study will undergo NavX CPM recording of the heart using the EnSite NavX Mapping system during the implantation of a cardiac resynchronization therapy device.

ELIGIBILITY:
Inclusion Criteria:

* Be undergoing a new St. Jude Medical CRT-D or CRT-P device implantation
* Have the ability to provide informed consent for study participation and be willing to comply with the prescribed perioperative evaluations

Exclusion Criteria:

* Have a recent myocardial infarction within 40 days prior to enrollment
* Have undergone cardiac surgery or coronary revascularization procedure within 3 months prior to enrollment or be scheduled for such procedures
* Be less than 18 years of age
* Be pregnant women
* Be currently participating in a clinical study that includes an active treatment arm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for implantation of a CRT pulse generator
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2007-12; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Sperzel, MD, Principal Investigator — Kerckhoff Klinik GmbH; Andre d'Avila, MD, Principal Investigator — Massachusetts General Hospital; Imran Niazi, MD, Principal Investigator — Arrhythmia Center of Southern Wisconsin, Ltd
Locations (1):
- St. Jude Medical, Sunnyvale, California, United States

REFERENCES:
- [Derived] Sperzel J, Brandt R, Hou W, Doelger A, Zdarek J, Rosenberg SP, Ryu K, Koh S, Yang M. Intraoperative characterization of interventricular mechanical dyssynchrony using electroanatomic mapping system--a feasibility study. J Interv Card Electrophysiol. 2012 Nov;35(2):189-96. doi: 10.1007/s10840-012-9695-0. Epub 2012 Jun 14. PMID 22695763